CLINICAL TRIAL: NCT05388266
Title: Effect of Paratracheal Pressure on Mask Ventilation in Anesthetized Obese Patients
Brief Title: Effect of Paratracheal Pressure on Mask Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 05112022
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paratracheal pressure (Experimental): After the induction of anesthesia, paratracheal pressure is applied during mask ventilation.
  Interventions: Other: Mask ventilation
- No pressure (Active Comparator): After the induction of anesthesia, no pressure is applied during mask ventilation.
  Interventions: Other: Mask ventilation

INTERVENTIONS:
Other: Mask ventilation — Mask ventilation is performed under paratracheal pressure or no pressure in a randomized, crossover manner.

SUMMARY:
This study aims to evaluate the effect of paratracheal pressure on mask ventilation in anesthetized obese patients in terms of expiratory tidal volume, and peak inspiratory pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a body mass index ≥ 30 kg.m-2 undergoing general anesthesia for elective surgery

Exclusion Criteria:

* Structural abnormalities or diseases in the face, neck, upper airway, or esophagus
* Increased risk of aspiration (pregnancy)
* Carotid artery stenosis, cerebrovascular disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Expiratory tidal volume | For 2 min of mask ventilation after the induction of anesthesia
  Volume controlled mechanical ventilation is delivered during mask ventilation. Expiratory tidal volumes on the monitor screen are recorded during mask ventilation

SECONDARY OUTCOMES:
Peak inspiratory pressure | For 2 min of mask ventilation after the induction of anesthesia
  Peak inspiratory pressure on the screen is recorded during mask ventilation.
Inadequate tidal volume | For 2 min of mask ventilation after the induction of anesthesia
  Incidence of tidal volume less than 150 mL is recorded.
Incidence of hypoxia | For 2 min of mask ventilation after the induction of anesthesia
  Occurrence of hypoxia (SpO2 <90%) is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Seol T, Kim H, Chang JE, Kang Y, Hwang JY. Effect of paratracheal pressure on the effectiveness of mask ventilation in obese anesthetized patients: a randomized, cross-over study. J Clin Monit Comput. 2024 Feb;38(1):31-36. doi: 10.1007/s10877-023-01048-8. Epub 2023 Jul 7. PMID 37418060